CLINICAL TRIAL: NCT04692363
Title: Prevention of Rituximab Related Flare by Plasmapheresis in Cryoglobulinemic Vascularitis
Brief Title: Plasmapheresis Before Rituximab in Cryoglobulinemia
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Other Study IDs: RECHMPL20_0683
Record Dates: First submitted 2020-12-30; First posted 2020-12-31 (Actual); Last update posted 2020-12-31 (Actual); Status verified 2020-12

CONDITIONS: Cryoglobulinemic Vasculitis
Keywords: Cryoglobulinemic vasculitis requiring rituximab therapy
MeSH Terms: conditions — Cryoglobulinemia, Familial Mixed

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Initial worsening following initiation of rituximab therapy in patients with cryoglobulinemic vasculitis was described in 3.6% of cases. This worsening is often a serious condition, with high levels of mortality.

The objective of our study is to evaluate the efficacy of preventive plasmapheresis prior to the introduction of rituximab performed in Montpellier France since 2013 by assessing the frequency and severity of this flare effect in these patients compared to those reported in the literature.

ELIGIBILITY:
Inclusion criteria:

* cryoglobulinemic vasculitis requiring rituximab treatment
* Patient ≥18 years old

Exclusion Criteria:

* Patient who reject the study protocol
* Patient < 18 years old

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patient with cryoglobulinemic vasculitis requiring rituximab treatment
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 1999-01-01 (Actual); Primary Completion 2021-12-01 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
comparison of frequency of occurrence of flare effects | 1 day
  comparison of frequency of occurrence of flare effects between patients who received plasmapheresis prior to rituximab compared to patients who did not.

SECONDARY OUTCOMES:
evaluation of the severity of the flare effect | 1 day
  evaluation of the severity of the flare effect
impact of known risk factors | 1 day
  investigation of the impact of known risk factors for this effect
evaluation of the safety of plasmapheresis in this indication | 1 day
  evaluation of the safety of plasmapheresis in this indication
evaluation of the efficacy of plasmapheresis on biological parameters | 1 day
  evaluation of the efficacy of plasmapheresis on biological parameters

CONTACTS AND LOCATIONS:
Overall Officials: Charles HERBAUX, assistant Professor, Study Director — University Hospital, Montpellier
Locations (1):
- Uhmontpellier, Montpellier, France

IPD SHARING:
Plan to Share IPD: Undecided
NC